CLINICAL TRIAL: NCT04305366
Title: MicroRNA Markers in Head and Neck Cancers
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12-1328.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-02-06; First posted 2020-03-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fine needle aspiration biopsy, blood, and saliva specimens. DNA will be isolated from tissue samples obtained and this DNA will be treated with Bisulfite and we will use the SBYR Green Florescent labeling system in conjunction with real-time quantitative PCR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancers: This study will target patients with a diagnosis squamous cell carcinoma in the head and neck. In addition, this study will also target patients undergoing tonsillectomy or sleep surgery as the control group. This study will aim to enroll an equal number of patients into both the study group and control group. However, this will be dependent on patient encounters within the adult ENT clinic.
  Interventions: Other: Tissue collection

INTERVENTIONS:
Other: Tissue collection — Blood draw, Fine Needle Aspiration, Saliva Swab, Tumor/tissue sample

SUMMARY:
The purpose of this study is to investigate the presence of miRNA markers in saliva, blood, FNA and tissue specimens in patients with and without head and neck cancer and evaluate whether these miRNA markers can provide prognostic or diagnostic clinical significance in the treatment of head and neck cancer patients.

DETAILED DESCRIPTION:
Micro RNA (miRNA) markers were initially discovered in 1993 and recent research has shown that they have great potential for use as both surveillance and prognostic markers in cancer treatment, as well as potential targets for cancer therapy. Recent research has identified several miRNA markers which appear to be potential markers for head and neck squamous cell carcinoma, and these have been tested in both mouse and human banked tumor samples. These investigators hypothesize that these markers may also be present in other tissues, including fine needle aspiration biopsy, blood, and saliva specimens, and will be sensitive and specific to patients with known head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 18 and 100
2. Patients who are seen and evaluated by a provider within the adult ENT clinic at University of Colorado Hospital
3. Patients that present with a current or past diagnosis of head and neck cancer -OR-Patients undergoing tonsillectomy or sleep surgery as standard of care (control group)

Exclusion Criteria:

1. Under the age of 18 or over the age of 100
2. Unwilling to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 500 patients will be enrolled in this study. Subjects to be enrolled in this study will already have a clinical relationship with a professional in the adult ENT clinic at University of Colorado Hospital.
  This study will target patients with a diagnosis squamous cell carcinoma in the head and neck. In addition, this study will also target patients undergoing tonsillectomy or sleep surgery as the control group. This study will aim to enroll an equal number of patients into both the study group and control group. However, this will be dependent on patient encounters within the adult ENT clinic.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Investigate the miRNA signature of samples | 5 years
  Tissue samples will be obtained and DNA will be isolated from those samples. DNA will be treated with Bisulfite and labelled with SBYR Green Florescent labeling system, in conjunction with real-time quantitative PCR for analysis. miRNA biomarkers idenfitied through PCR will be collected.
Develop biomarkers from fine needle aspiration biopsies and other specimens, using real-time PCR, for surveillance of HNSCC patients. | 5 years
  Fine needle aspiration (FNA) biopsies, saliva, serum and tumor samples will be collected from HNSCC patients and controls. Samples will undergo real-time PCR using miRNA biomarkers. The efficacy of these biomarkers will be collected, to determine the status of the Head/Neck Cancer as the study progresses

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Long Lu, MD PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No